CLINICAL TRIAL: NCT03002805
Title: A Phase I Trial of CBT-1® in Combination With Doxorubicin in Patients With Locally Advanced or Metastatic, Unresectable Sarcomas Previously to Have Progressed on 150 mg/m2 or Less of Doxorubicin
Brief Title: CBT-1® in Combination With Doxorubicin in Patients With Metastatic, Unresectable Sarcomas Who Previously Progressed on Doxorubicin
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CBA Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STS-1701
Record Dates: First submitted 2016-12-15; First posted 2016-12-26 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Sarcoma
Keywords: Phase I; CBT-1®; Doxorubicin; Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: CBT-1® — CBT-1®, oral, on days 1-7 of each cycle 21-day cycle. Participants will be assigned to dose level of CBT-1®:
  Dose level 1 - 50 mg/m2/day Dose level 2 - 100 mg/m2/day Dose level 3 - 150 mg/m2/day Dose level 4 - 200 mg/m2/day Dose level 5 - 250 mg/m2/day Dose level 6 - 300 mg/m2/day doxorubicin, 37.5 mg/m2, IV, on days 5 and 6 of each cycle Study treatment discontinued after 450 mg/m2 lifetime cumulative dose of doxorubicin reached or after 4-5 cycles completed.
  Other Names: doxorubicin

SUMMARY:
This study evaluates the combination of CBT-1® and doxorubicin for the treatment of metastatic, unresectable sarcoma in patients who have progressed after treatment with 150mg/m2 or less of doxorubicin. Participants will receive CBT-1® on days 1-7 of each 21-day cycle, as well as doxorubicin on days 5 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Locally advanced or metastatic, unresectable sarcoma that has progressed after treatment with 150 mg/m2 or less of doxorubicin or anthracycline equivalent
* Measurable disease by RECIST 1.1
* ECOG performance status of ≤ 1
* Life expectancy of > 3 months
* Able to swallow pills
* Adequate bone marrow and organ function as defined as:
* Hemoglobin > 9 g/dl
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin < 1.5 X ULN
* AST(SGOT)/ALT(SGPT) ≤3 X ULN (including patients with liver metastases)
* Creatinine <1.5 X ULN
* Cardiac ejection fraction >50% (by echocardiogram or MUGA) within 15 days of enrollment
* Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to enrollment.
* Participants must be willing and able to comply with the study scheduled visits, laboratory tests, and other procedures outlined in the protocol.
* Pre-menopausal women must have a negative pregnancy test before study entry. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for at least six weeks after treatment discontinuation. Acceptable methods of contraception include intrauterine device (IUD), oral contraceptive, subdermal implant, double barrier and/or complete abstinence (non-periodic).
* Washout period prior to Day 1 Cycle 1:
* 3 weeks since last chemotherapy or therapeutic radiation therapy
* 4 weeks or 3 half-lives since prior antibody-based therapy, whichever is shorter
* 2 weeks since any oral anti-neoplastic or oral investigational agent
* Resolution of treatment-related toxicity to < grade 1; alopecia and cutaneous toxicity are allowed < grade 2
* >1 week since palliative RT
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior exposure to CBT-1
* Previously untreated sarcomas
* Low-grade sarcomas as well as alveolar soft parts sarcoma, clear cell sarcoma, extraskeletal myxoid chondrosarcoma, well-differentiated liposarcoma, gastrointestinal stromal tumor, chordoma
* Participants receiving other investigational agents
* Participants with known uncontrolled brain metastases
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, chronic indwelling drains, history of interstitial pneumonitis or pulmonary fibrosis or psychiatric illness/social situations that would limit compliance with study requirements
* Actively breastfeeding women unless it is interrupted during treatment and at least 6 weeks after treatment discontinuation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of CBT-1® when combined with doxorubicin | 3 years

SECONDARY OUTCOMES:
Recommended phase 2 dose (RP2D) of CBT-1® when combined with doxorubicin | 3 years
Disease Control Rate (DCR) of CBT-1® when combined with doxorubicin | week 12
  DCR = Overall Response Rate [ORR = Complete Response + Partial Response] + Stable Disease by RECIST 1.1
Overall Response Rate | 3 years

OTHER OUTCOMES:
Correlation of DCR, ORR and PFS to disease subtype | 3 years
Correlation of P-gp expression at baseline to P-gp expression after treatment | 3 years
Correlation of tumor response to P-gp inhibition by CBT-1® | 3 years
Presence of CBT-1® in tumor tissue | 3 years

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Mayo Clinic, Jacksonville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903